CLINICAL TRIAL: NCT03121287
Title: Early Imaging Biomarkers to Predict Radiation-Induced Cardiopulmonary Toxicity in Patients With Thoracic Malignancies
Brief Title: Early Imaging Biomarkers in NSCLC
Status: Completed | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: UMCC 2015.006; HUM00097162 (Other: U-M IRB)
Record Dates: First submitted 2017-04-14; First posted 2017-04-20 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Thoracic Cancer
MeSH Terms: interventions — X-Rays; Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lung or Esophageal Patients: Patients with lung or esophageal cancer undergoing conventionally-fractionated radiation therapy. Interventions to be administered include: Imaging Biomarkers using Volumetric CT Scans, Pulmonary using Pulmonary Function Test & 6Minute Hall Walk, Imaging using Cardiac MRI, Specimen Collection using Blood Draws.
  Interventions: Other: Imaging Biomarkers; Other: Pulmonary; Other: Imaging; Other: Specimen Collection

INTERVENTIONS:
Other: Imaging Biomarkers — Whole lung volumetric CT scans
Other: Pulmonary — Pulmonary Function Tests & 6 minute hall walk
Other: Imaging — Cardiac MRI
Other: Specimen Collection — Blood draw

SUMMARY:
The purpose of this study is to investigate if cardiac MRI, blood biomarkers, and lung CT scans can detect early changes to the associated with radiation therapy in patients receiving radiation treatment for thoracic cancer.

DETAILED DESCRIPTION:
This study seeks to investigate the utility of novel imaging biomarkers, namely whole lung volumetric CT scans and cardiac MRI, to non-invasively identify early pathologic changes in pulmonary and cardiac function resulting from thoracic radiation. The ability to identify these changes during the course of treatment offers a powerful tool to optimize radiation dose distributions within uninvolved normal tissue by adapting treatment to the individual patient response. In addition it may lead to other therapeutic interventions designed to reduce long term cardiopulmonary toxicity.

The cardiac MRI will be performed using Aminophylline, Gadopentetate Dimeglumine and Regadenoson. These are not FDA approved for this purpose, but are being used off label and are IND exempt. Additionally, patients will be consented with an optional choice to retain research blood samples for 15 years after the completion of the study. This will allow cutting edge analysis for biomarkers that may be discovered in the future.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving once daily fractionated intrathoracic radiation therapy for:
* Stage IIA-IIIB non-small cell lung cancer
* Limited stage small cell lung cancer
* Stage I-III esophageal cancer (neoadjuvant or definitive)
* Patients must be 18 years of age or older
* Must not be claustrophobic
* Must have adequate kidney function

Exclusion Criteria:

* Patients with small cell lung cancer receiving twice daily (b.i.d.) radiation
* Patients with esophageal cancer receiving trastuzamab
* Pregnancy or lactation
* Claustrophobia
* Inability to lie flat for 60-90 minutes
* Renal dysfunction with eGFR <60 mL/min/1.73 m2
* Allergy to gadolinium containing contrast media
* Implanted devices, metallic hazards or other conditions presenting a contraindication to 3Tesla cardiac MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing conventionally-fractionated intrathoracic radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2015-09-23 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Lung Function | 1 Year post treatment
  To characterize longitudinal changes in lung function using a voxel-wise image analysis technique of whole-lung CT scans in patients undergoing intrathoracic radiation therapy.

SECONDARY OUTCOMES:
Change from Baseline in Myocardial Tissue | 1 Year post treatment
  To assess longitudinal changes in myocardial tissue and coronary vasculature physiology, using cardiac MR in patients undergoing intrathoracic radiation therapy.
Change from Baseline in Myocardial Tissue | 1 Year post treatment
  To assess longitudinal changes in myocardial tissue and coronary vasculature physiology, including microvascular dysfunction, using cardiac MR in patients undergoing intrathoracic radiation therapy.
Change from Baseline in Myocardial Tissue | 1 Year post treatment
  To assess longitudinal changes in myocardial tissue and coronary vasculature physiology, including diffuse fibrosis, using cardiac MR in patients undergoing intrathoracic radiation therapy.
Radiation Predictors from Baseline in Cardiopulmonary Changes | 1 Year post treatment
  To explore radiation dosimetric predictors of CT- and MR-detectible cardiopulmonary changes.

OTHER OUTCOMES:
Radiation Induced Change from Baseline in Imaging | 6 month and 1 year post treatment
  To determine if early imaging-based changes are associated with radiation induced pulmonary and cardiac injury at 6- and 12-months

CONTACTS AND LOCATIONS:
Overall Officials: Shruti Jolly, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No